CLINICAL TRIAL: NCT06593028
Title: Feasibility of a Pilot Intervention Designed to Increase SNAP Fruit and Vegetable Incentive Program Use for Families With Food Insecurity
Brief Title: Feasibility of Strategies to Increase SNAP Fruit and Vegetable Incentive Program Use for Families With Food Insecurity
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of South Carolina (Other)
Responsible Party: Principal Investigator, Elizabeth Adams, Assistant Professor, University of South Carolina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Pro00120539
Record Dates: First submitted 2024-09-06; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Dietary Habits
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Veggie Vouchers pilot intervention (Experimental): During well-child visits, caregivers received brief education from pediatricians about a Supplemental Nutrition Assistance Program (SNAP) fruit and vegetable incentive program in South Carolina. Following the clinic visit, a free trial for this SNAP fruit and vegetable incentive program was then offered. The free trial consisted of 3 vouchers, each good for one free fruit and vegetable box.
  Interventions: Behavioral: Veggie Vouchers pilot

INTERVENTIONS:
Behavioral: Veggie Vouchers pilot — This intervention aims to increase awareness and use of a Supplemental Nutrition Assistance Program (SNAP) fruit and vegetable incentive program in South Carolina among families with young children experiencing food insecurity. To do so, brief education about this SNAP program is delivered by pediatricians to caregivers during well-child visits. Subsequently, caregivers are given 3 free produce boxes as a free trial of this program to incentivize first time use.

SUMMARY:
The Veggie Vouchers pilot intervention aimed to increase awareness and utilization of an existing SNAP F&V incentive program in South Carolina for families with food insecurity. Social determinants of health screenings were leveraged in a pediatric clinic to identify eligible families and provide information about this program. A free trial was then offered, with the long-term goal of increasing program use after the free trial ended. The primary aim was feasibility and acceptability of the Veggie Vouchers intervention among pediatricians and families.

ELIGIBILITY:
Caregiver Inclusion Criteria:

* 18 years of age or older
* Had a child 2-17 years of age
* Child lived in their home 50% of the time or more
* Child was a patient of the general pediatrics clinic enrolled in this study
* English-speaking
* Enrolled in SNAP
* Experiencing household food insecurity

Caregiver Exclusion Criteria:

* Had purchased fruits and vegetables within the past year at the community food site participating in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Intervention feasibility: recruitment screening eligibility | Through study completion, approximately 1 year
  Percent of caregivers screened who were eligible
Intervention feasibility: recruitment screening enrollment | Through study completion, an average of 1 year
  Percent of eligible caregivers who enrolled
Intervention feasibility: recruitment duration | Through study completion, an average of 1 year
  Duration to reach the target sample
Intervention feasibility: retention attendance | Through study completion, an average of 1 year
  Assessment completion rates
Intervention feasibility: retention dropout | Through study completion, an average of 1 year
  Percent of sample that drops out or is lost to follow-up
Intervention acceptability: caregivers | Upon completing the intervention, approximately 5 months after baseline
  Acceptability was assessed via surveys on caregivers satisfaction of the intervention
Intervention acceptability: pediatricians | Upon completing the intervention, approximately 1 year
  Acceptability was assessed via surveys on pediatricians perceptions of the intervention
Intervention acceptability | Upon completing the intervention, approximately 3 months after baseline
  Exit surveys were used to assess reasons for low utilization of the intervention
Intervention utilization: free trial redemption | Through free trial period, approximately 3 months from baseline
  How many free trial vouchers were ordered and received
Intervention utilization: SNAP purchases (box frequency) | Through study completion, approximately 1 year
  Number of additional fruit and vegetable boxes purchased using SNAP electronics benefit card
Intervention utilization: SNAP purchases (family uptake) | Through study completion, approximately 1 year
  How many families purchased additional fruit and vegetable boxes using their SNAP electronics benefit card

SECONDARY OUTCOMES:
Household food insecurity | Baseline, after receiving each free fruit and vegetable box (~1x/month for 3 months after baseline), and end of the intervention (~5 months after baseline for redeemers; 3 months after baseline for non-redeemers)
  The 18-item United States Department of Agriculture (USDA) Household Food Security Module was used to assess household food security status. Scores range 0 to 18. Higher scores indicate greater degrees of food insecurity.
Household nutrition security | Baseline, after receiving each free fruit and vegetable box (~1x/month for 3 months after baseline), and end of the intervention (~5 months after baseline for redeemers; 3 months after baseline for non-redeemers)
  The Household Nutrition Security scale was used to assess a household's ability to acquire foods that meet their nutritional needs without resource limitations or worry. Scores range 0 to 4. Higher scores indicate a greater degree of household nutrition security.
Household healthfulness choice | Baseline, after receiving each free fruit and vegetable box (~1x/month for 3 months after baseline), and end of the intervention (~5 months after baseline for redeemers; 3 months after baseline for non-redeemers)
  The Household Nutrition Security scale was used to assess a household's ability to acquire foods that meet their health needs without resource limitations or worry. Scores range 0 to 4. Higher scores indicate a greater degree of household healthfulness choice.
Household dietary choice | Baseline, after receiving each free fruit and vegetable box (~1x/month for 3 months after baseline), and end of the intervention (~5 months after baseline for redeemers; 3 months after baseline for non-redeemers)
  The Household Dietary Choice scale was used to assess a household's ability to acquire foods that meet their dietary preferences without resource limitations or worry. Scores range 0 to 4. Higher scores indicate a greater degree of household dietary choice
Dietary intake | Baseline, after receiving each free fruit and vegetable box (~1x/month for 3 months after baseline), and end of the intervention (~5 months after baseline for redeemers; 3 months after baseline for non-redeemers)
  The National Cancer Institute's Dietary Screener Questionnaire (DSQ) was used to assess caregiver's report of children's dietary intake. Responses are quantified as cup equivalents per day, grams per day, milligrams per day, ounce equivalents per day, or teaspoon equivalents per day. Whether higher or lower numbers indicate more healthful or less healthful dietary intake is specific to each nutrient.

CONTACTS AND LOCATIONS:
Locations (1):
- University of South Carolina, Columbia, South Carolina, United States

REFERENCES:
- [Derived] Adams EL, Savidge M, Reesor-Oyer L, Draper C, Steeves EA, Bean MK, Figueroa R, Stephenson K, Weaver RG, Armstrong B, Beets M, Burkart S. The Veggie Vouchers intervention to promote SNAP fruit and vegetable incentive program use for families with food insecurity: a single arm feasibility study. Pilot Feasibility Stud. 2025 Dec 2;11(1):157. doi: 10.1186/s40814-025-01732-3. PMID 41331706